CLINICAL TRIAL: NCT05580887
Title: Intestinal Microbiota Impact for Prognosis and Treatment Outcomes in Early Luminal Breast Cancer and Pancreatic Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Moscow Clinical Scientific Center (Other)
Responsible Party: Sponsor
Other Study IDs: Microbiome_BC&PnC
Record Dates: First submitted 2022-06-21; First posted 2022-10-14 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Breast Cancer; Pancreas Cancer
MeSH Terms: conditions — Breast Neoplasms; Pancreatic Neoplasms | interventions — Doxorubicin; Cyclophosphamide; Paclitaxel; Carboplatin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with luminal A breast cancer
- Patients with high risk luminal B breast cancer
  Interventions: Drug: Doxorubicin; Drug: Cyclophosphamid; Drug: Paclitaxel; Drug: Carboplatin
- Patients with high pancreatic cancer
  Interventions: Drug: mFOLFIRINOX

INTERVENTIONS:
Drug: mFOLFIRINOX — every 2 weeks: Oxaliplatin 65 mg/m2 IV over 3 hours on Day 1 Irinotecan 150 mg/m2 IV over 90 minutes on Day 1 Leucovorin(l-LV) 200 mg/m2 IV over 2 hours on Day 1 5-Fluorouracil 2.4 g/m2 for 46 hours continuous infusion.
  Groups: Patients with high pancreatic cancer
Drug: Doxorubicin — dose dense doxorubicin and cyclophosphamide (AC) x 4 every 2 weeks followed by 12 weekly PAClitaxel + CARBOplatin every 21 days for 4 cycles
  Groups: Patients with high risk luminal B breast cancer
Drug: Cyclophosphamid — dose dense doxorubicin and cyclophosphamide (AC) x 4 every 2 weeks followed by 12 weekly PAClitaxel + CARBOplatin every 21 days for 4 cycles
  Groups: Patients with high risk luminal B breast cancer
Drug: Paclitaxel — dose dense doxorubicin and cyclophosphamide (AC) x 4 every 2 weeks followed by 12 weekly PAClitaxel + CARBOplatin every 21 days for 4 cycles
  Groups: Patients with high risk luminal B breast cancer
Drug: Carboplatin — dose dense doxorubicin and cyclophosphamide (AC) x 4 every 2 weeks followed by 12 weekly PAClitaxel + CARBOplatin every 21 days for 4 cycles
  Groups: Patients with high risk luminal B breast cancer

SUMMARY:
The gut microbiota (GM) can influence as effectiveness of immunotherapy as prognosis factor in cancer patients. The goal of the study to identify GM pattern is associated with poor and favourable treatment outcomes in breast cancer and pancreatic cancer patients for further treatment strategy proper planning.

ELIGIBILITY:
Inclusion Criteria:

* untreated early HR+ HER2- BC:

  1. planned neoadjuvant chemotherapy: dose dense doxorubicin and cyclophosphamide (AC) x 4 every 2 weeks followed by 12 weekly PAClitaxel + CARBOplatin every 21 days for 4 cycles
  2. TanyN1-3M0 Ki67>40% G3
  3. ECOG 0-1
* untreated early HR+ HER2- BC:

  1. TanyN0M0 Ki67<20% G1
  2. ECOG 0-1
  3. planned induction endocrine therapy (letrozole/anastrazole/tamoxifen)
* untreated locally-advanced and/or borderline resectable pancreas cancer:

  1. planned (neo)adjuvant chemotherapy: mFOLFIRINOX
  2. previous surgery ( only R0 resection) is allowed
  3. ECOG 0-1
  4. histology diagnosis verification
* Informed consent
* Eligible blood&fecal samples and tumor tissue for different time points

Exclusion Criteria:

* autoimmune disease
* active steroid therapy
* ECOG > 2
* any previous therapy for breast cancer
* metastatic cancer
* antibiotic use less than 28 days
* other tumor

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Early lum A and high risk lum B HER2- breast cancer
  * Locally advanced resectable and/or borderline resectable panreatic cancer
Sampling Method: Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2022-05-12 (Actual); Primary Completion 2025-05-12 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Intestinal bacterial structure in BC and PnC (separately) patients with disease progression | 24 months
  Intestinal bacterial structure will performed by 16S RNA gene sequencing

SECONDARY OUTCOMES:
Change from baseline of ctDNA level in the each type of breast cancer patients from diagnosis till 24 months after completion neoadjuvant chemotherapy followed by surgery | 30 months (6 months treatment period+24 months follow up)
  Change from baseline of ctDNA level in the each type of breast cancer patients from diagnosis till 24 months after completion neoadjuvant chemotherapy followed by surgery
Change from baseline in intestinal bacterial structure in patients with early high risk luminal breast cancer of recurrence and increasing ctDNA level who are receiving neo/adjuvant chemotherapy regimens | 30 months
  Change from baseline in intestinal bacterial structure in patients with early high risk luminal breast cancer of recurrence and increasing ctDNA level who are receiving neo/adjuvant chemotherapy regimens.
  Intestinal bacterial structure will performed by 16S RNA gene sequencing.
Change from baseline in intestinal bacterial structure in PnC patients 12 months after after the completion of combined treatment | 18 months (6 months treatment period+ 12 months follow up)
  Intestinal bacterial structure will performed by 16S RNA gene sequencing
Change from baseline in intestinal bacterial structure in PnC patients with disease relapse on or after combined treatment completion (follow up 12 months) | 18 months (6 months treatment period+ 12 months follow up)
  Intestinal bacterial structure will performed by 16S RNA gene sequencing

CONTACTS AND LOCATIONS:
Locations (1):
- Moscow Clinical Scientific Center named after AS Loginov, Moscow, Not Required, Russia